CLINICAL TRIAL: NCT06107075
Title: Investigating the Effects of Dietary Phospholipids on Measures of Human Brain Health and Psychological Wellbeing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Volac International Ltd (Unknown)
Responsible Party: Principal Investigator, Philippa Jackson, Principal Investigator, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 66CH1
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Mood; Cognitive Change; Well-Being, Psychological
Keywords: Cognition; Mood; Well-being; Physical Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomised, placebo-controlled, double-blind, parallel groups design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor)- Treatment will be blinded according to the randomisation schedule by a researcher who has no other involvement in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioactive whey protein concentrate containing phospholipids (Experimental): Bioactive whey protein concentrate containing phospholipids 40g powder mixed with 350ml water consumed once daily for 12 weeks alongside their fattiest meal of the day.
  Interventions: Dietary Supplement: Active
- Placebo (Placebo Comparator): Placebo powder matched for macronutrient and caloric content containing pea protein around 40g powder mixed with 350ml water consumed once daily for 12 weeks alongside their fattiest meal of the day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Active — 40g bio-active whey protein concentrate powder containing phospholipids
  Other Names: active treatment
  Arms: Bioactive whey protein concentrate containing phospholipids
Dietary Supplement: Placebo — around 40g pea protein powder not containing phospholipids
  Other Names: Placebo Treatment
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the effects of 6- and 12-week supplementation of a bioactive whey protein concentrate drink containing dairy phospholipids on cognitive function and mood in healthy young to middle aged adults.

The proposed randomised, double blind, placebo-controlled, parallel groups design methodology will assess the cognitive, mood and lifestyle effects of 40g per day of bioactive whey protein concentrate powder mixed with water and matched placebo prior to (baseline) and after -6 and 12-week supplementation. The trial will utilise the COMPASS cognitive assessment system (Northumbria University) during the laboratory visits to measure performance on the cognitive tasks and a range of mood measures between visits examining general mood, stress, depression, anxiety, sleep quality, fatigue, and physical symptoms.

Additionally, dairy dietary habits will be recorded throughout to allow for any significant changes to diet to be assessed for the potential influence on the outcome variables.

Participants will be asked not to make any major changes to their diet or exercise regime for the duration of the trial. This will be checked by asking the participant if there has been any significant changes at each visit.

Blood samples will also be taken from a subset of participants who opt into this part of the trial to measure any changes to plasma phospholipid profiles.

220 participants will participate, aged 25-49, and self-report as in good health. Participants will be supplied with the treatment whilst visiting the research centre on testing days and will then consume treatment at home daily. Participants will record the time they take their treatment each day in a diary that will then be returned to the research team at the end of the study testing period.

DETAILED DESCRIPTION:
The study will follow a randomised, placebo-controlled, double-blind, parallel groups design.

Participants will attend the research centre on four separate occasions, which will include a screening/training visit, pre intervention testing visit, a mid-point testing visit (at 6 weeks), and a completion of intervention testing visit (at 12 weeks). There will be 5 appointments in total including the online appointment to check for eligibility. The remote screening session will be completed via telephone call and will comprise briefing on the requirements for the study, answering any initial questions, obtaining of informed consent via completion of an online consent form, health screening, collection of demographic information, and completion of the Caffeine Consumption Questionnaire (CCQ).

The introductory/training visit to the laboratory will begin with physiological eligibility measures that cannot be completed remotely (e.g., blood pressure, height and weight, waist-to-hip ratio) followed by training on the cognitive and mood measures.

Opportunity sampling will be used to recruit participants. The study will include 220 healthy participants aged between 25-49 years, who will receive 12 weeks' worth of either 40g per day of bioactive whey protein concentrate powder containing dairy phospholipids (to be mixed with approx. 350ml water to form a drink), or similar amount per day of matched placebo powder. Participants will be randomly allocated to either the treatment or placebo group and neither the participant nor the researcher will know which group they have been allocated to. Full instructions of how and when to take treatment each day will be explained to the participants when treatment is provided at testing visit 1.

The day before each of the study testing days, participants will be sent a link to a set of questionnaires they must complete before attending the lab on the following day. The set includes questionnaires measuring perceived stress, sleep quality, levels of fatigue, physical symptoms, and general health and well-being. The questionnaires should take the participants approx. 45 minutes to complete on their computer, smartphone, or tablet at home.

On each of the three study testing days (Day 1, 42, and 84) participants will attend the research centre, having abstained from alcohol for 24 hours, and caffeine overnight, following a standardised breakfast of cereal and/or toast at home no later than 1 hour prior to arrival. Upon arrival to the research centre, participants continued eligibility will be checked before completing the 1 hour long computerised cognitive assessment using the Computerised mental performance assessment system (COMPASS). The cognitive assessment will employ a broad selection of tasks assessing performance within the "Attention", "Working Memory", "Episodic Memory", "learning" and "Executive Function" cognitive domains. The cognitive demand battery (CDB), which assess cognitive functioning and subjective mental fatigue during sustained performance of mentally demanding tasks, will also be incorporated. Upon completion of the computerised cognitive assessment, participants will complete the NASA task load index (NASA TLX) to measure perceived task mental demand.

Participants will additionally complete a treatment guess form at their final visit and will be fully debriefed.

Participants that opt into the blood sampling portion of this study will also attend the research centre on two separate additional occasions, the day (or two days) before the first and final testing visit, to have their blood taken. Participants will be required to attend the research centre fasted and therefore all blood draw appointments will be held in the morning. A venous blood sample will be taken by a trained phlebotomist. Samples will then be processed and stored at Northumbria University until time of analysis where they will be analysed for plasma phospholipid profiles. These additional blood visit will last approx. 15 minutes per visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants must self-assess themselves as being in good health.
* Participants must be aged 25 to 49 years at the time of giving consent.
* Participant must be fluent in English and/or English is their first language

Exclusion Criteria:

* Have any pre-existing medical conditions/illness which will impact taking part in the study. There may be other, unforeseen exceptions and these will be considered on a case-by-case basis: i.e., participants may be allowed to progress to screening if they have a condition/illness which would not interact with the active treatments or impede performance. It is therefore worth discussing any medical conditions with the researcher prior to booking lab appointments
* Are currently taking any prescription medications (NOTE the explicit exceptions to this are contraceptive treatments for female participants, and those taking "as needed" in the treatment of asthma and/or hay fever. There may be other instances of medication use which, where no interaction with the active treatment is likely, and which would not be expected to have any impact on brain function, participants may be able to progress to screening
* Have high blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg). NOTE: that we must measure this in the lab using our blood pressure monitors and can only use our measurements to assess eligibility rather than home or GP readings
* Have a Body Mass Index (BMI) outside of the range 18.5-35 kg/m2.
* Are pregnant, seeking to become pregnant or lactating.
* Have been diagnosed with a neurological condition, or assessed as having a learning/behavioural or neurodevelopmental difference (e.g. dyslexia, autism, ADHD.
* Have a visual impairment that cannot be corrected with glasses or contact lenses (including colour-blindness)
* Smoke tobacco or vape nicotine or use nicotine replacement products (if you have recently quit smoking or using replacements you must have stopped using them altogether for a period of 3 months before participating in this study)
* Have excessive caffeine intake (>500 mg per day). Note: This will be calculated at screening but feel free to query this with the researcher prior to attendance
* Have relevant food allergies/ intolerances/ sensitivities
* Have taken antibiotics within the past 4 weeks.
* Have taken dietary supplements e.g., vitamins, omega 3 fish oils etc. in the last 4 weeks (Note: participation is possible following a 4 week supplement wash out prior to participating and for the duration of the study on the proviso that the supplements they are taking are out of choice and not medically prescribed or advised. Please discuss with the researcher if unsure. NOTE: we would never advise stopping supplements prescribed by your doctor e.g., iron, calcium etc., only those you use out of choice)
* Have any health condition that would prevent fulfilment of the study requirements (this includes non-diagnosed conditions for which no medication may be taken)
* Are unable to complete all of the study assessments (this will be assessed by the researcher at your training appointment, you must be able to reach minimum scores for each of the cognitive tasks to progress with the trial)
* Are currently participating in other clinical or nutrition intervention studies, or have in the past 4 weeks
* Have been diagnosed with/ undergoing treatment for alcohol or drug abuse in the last 12 months.
* Have been diagnosed with/ undergoing treatment for a psychiatric disorder in the last 12 months, including a medical diagnosis of anxiety or depression.
* Suffers from frequent migraines that require medication (more than or equal to 1 per month)
* Have any sleep disorders or take any sleep medications.
* Have any known active infections.
* Have, previously have had, or think you are at risk of having syphilis, hepatitis, the Human T - lymphotropic virus or the Human Immunodeficiency Virus (HIV)
* Have ever had breast cancer and/or a mastectomy.
* Have haemophilia or any similar clotting/blood disorder.
* Have had unprotected sexual intercourse with any person from an HIV high risk population.
* Have ever been involved in intravenous drug use.
* Does not have a bank account (required for payment)
* Are non-compliant with regards treatment consumption
* Follow an "extreme" or very "strict" diet i.e., Keto, very high protein, sugar free, raw paleo etc.
* Are planning a major lifestyle change regarding diet or exercise regime in the next 3 months.
* Have a current diagnosis of renal impairments or phenylketonuria

Ages: 25 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive function - Cognitive domain factor score | prior to (baseline) and following chronic dose of intervention at 6 weeks and 12 weeks.
  Effects of supplementation on the cognitive domain memory, measured using the following tasks through the Computerised Mental Performance Assessment System (COMPASS, Northumbria University) :Numeric Working Memory, immediate word recall, delayed word recall, delayed word recognition, and delayed picture recognition. Participants will receive scores of accuracies on all tasks, which will be in the form of the percentage of responses correct. Higher scores indicate better memory performance, lower scores indicate worse memory performance.

SECONDARY OUTCOMES:
Profile of Mood States (POMS) | prior to (baseline) and following 6- and 12-week chronic intervention
  65-item measure, summed to create measures of vigour-activity (range 0-32), tension-anxiety (range 0-36), fatigue-inertia (0-28), depression-dejection (0-60), confusion-bewilderment (0-28), and anger-hostility (0-48). Higher scores indicate higher current levels of each aspect of mood. Answers are rated using a 5-point scale between "not at all (0)" and "extremely (4)".
Perceived Stress Scale (PSS) | prior to (baseline) and following 6- and 12-week chronic intervention
  10-item measure, summed to create a single value with higher scores indicating higher levels of stress. Scores can range from 0 to 40. Scores ranging from 0-13 would be considered low perceived stress, scores ranging from 14-26 would be considered moderate perceived stress, and scores ranging from 27-40 would be considered high perceived stress.
Perceived Stress Reactivity Scale (PSRS) | prior to (baseline) and following 6- and 12- week chronic intervention
  23-item measure, summed to create measures of prolonged reactivity (scores from 0-8), reactivity to work overload (scores from 0-10), reactivity to social conflict (scores from 0-10), reactivity to failure (scores from 0-8), reactivity to social evaluation (scores from 0-10), and perceived stress reactivity total (scores from 0-46). Higher scores indicate higher perceived stress reactivity.
The Cohen-Hoberman Inventory of Physical Symptoms (CHIPS) | Prior to (baseline) and following 6- and 12- week chronic intervention
  33-item measure, summed to create a measure of number of health complaints in the previous 2 weeks. Answers are recorded using a 5-item Likert scale ranging from 0 (meaning they have not been bothered by this problem), to 4 (meaning the problem has been an extreme bother). All the scores across the 33 items will be summed together to create a total score. The score will range from 0 to 132 and will indicate how extensively a participant has been bothered by physical symptoms in the previous 2-week period (higher scores indicating more bothered by physical symptoms).
Subjective sleep via the Patient-Reported Outcome Measurement, Information System Sleep Disturbance Scale- shoer form (PROMIS-SD) | prior to (baseline) and following 6- and 12-week chronic intervention
  prior to (baseline) and following 6- and 12-week chronic intervention Description: 8-item measure, summed to create a single value with higher scores indicating higher levels of sleep disturbances. Responses are recorded using a 5-item Likert scale ranging from 1 (Not at all) to 5 (Very much). Total score will therefore range from 8 to 40.
Depression, Anxiety and Stress Scale (DASS-21) | Prior to (baseline) and following 6- and 12-week chronic intervention
  21 item measure, summed to create 3 component scores; depression, anxiety and stress. Responses recorded using a 4-item Liker scale (0-3). Raw score range rom 0-63 as an indication of overall distress (the higher the score the more general distress). Depression, anxiety, and stress scored between 0 and 21. The higher the score indicated higher levels of depression, anxiety and stress.
Fatigue Assessment Scale (FAS) | prior to (baseline) and following 6- and 12- week chronic supplementation
  10-item measure, summed to create a measure of over perceived fatigue where less than 22 indicates "normal" levels of fatigue, 22-34 indicates mild-to-moderate fatigue and 35 or higher indicates severe fatigue. Total score ranges from 10 to 50.
Perceived task demand via the NASA Task Load Index (NASA TLX) | Following each of the cognitive assessments (3) at baseline, 6- weeks, and 12-week supplementation.
  five 7-point scales summed to create a measure of perceived mental workload of the cognitive tasks. Higher scores indicating higher perceived task demand.
Cognitive function- individual cognitive task score | prior to (baseline) and following 6- and 12- week chronic supplementation
  location learning task (accuracy), immediate word recall (accuracy), delayed word recall (accuracy) , delayed word recognition (accuracy and reaction time), delayed picture recognition (accuracy and reaction time), simple reaction time (reaction time), numeric working memory (accuracy and reaction time), Stroop (accuracy and reaction time), delayed location learning task (accuracy), and arrow flankers measured through the software Computerised Mental Performance Assessment System (COMPASS), Northumbria University. Scores for accuracy are the percentage of correct responses on that task. Reaction time is measures in milliseconds, and the lower the score the faster the response time.
Cognitive function- cognitively demanding tasks | prior to (baseline) and following 6- and 12- week supplementation
  cognitive function (scores based on number of answers correct within the time frame for serial subtractions, and accuracy of correct responses and reaction time measured in milliseconds for rapid visual information processing task) and mental fatigue (measured using a bespoke visual assessment scale) during extended performance of cognitively demanding tasks (cognitive demand battery, comprising serial 3s subtractions, serial 7s subtractions, rapid visual information processing task, and mental fatigue scales, repeated 3 times), measured though the software Computerised Mental Performance Assessment System (COMPASS), Northumbria University.
Changes to blood plasma phospholipid profiles | prior to (baseline) and following 12-week chronic supplementation
  Using venous blood samples to measure changes to plasma phospholipid profiles pre and post intervention.
Cognitive function - cognitive domain factor scores | prior to (baseline) and following chronic dose of intervention at 6 weeks and 12 weeks.
  Speed of attention (reaction time), accuracy of attention (accuracy), speed of memory (reaction time), accuracy of working memory (accuracy), accuracy of executive function (accuracy), learning (accuracy), delayed learning (accuracy) and accuracy of episodic memory (accuracy) measured by Computerised Mental Performance Assessment System (COMPASS, Northumbria University). Scores for accuracy are the percentage of correct responses on that task. Reaction time is measures in milliseconds, and the lower the score the faster the response time.

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University - Brain Performance and Nutrition Research Centre, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No